CLINICAL TRIAL: NCT02719028
Title: A Prospective, Double Blind, Randomized, Placebo-controlled Trial of Antroquinonol in Patients With Hypercholesterolemia and Hyperlipidemia
Brief Title: Trial of Antroquinonol in Patients With Hypercholesterolemia and Hyperlipidemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GHLIP-2-001
Record Dates: First submitted 2016-03-10; First posted 2016-03-25 (Estimated); Results first posted 2019-12-20 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Hyperlipidemias
MeSH Terms: conditions — Hyperlipidemias | interventions — antroquinonol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (antroquinnonol 50mg or Placebo) 3 capsules once a day.
  Interventions: Drug: placebo
- Antroquinonol 50 mg PO (Experimental): Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (antroquinnonol 50mg or Placebo) 3 capsules once a day.
  Interventions: Drug: Antroquinonol; Drug: placebo
- Antroquinonol 100 mg PO (Experimental): Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (antroquinnonol 50mg or Placebo) 3 capsules once a day.
  Interventions: Drug: Antroquinonol; Drug: placebo
- Antroquinonol 150 mg PO (Experimental): Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (antroquinnonol 50mg or Placebo) 3 capsules once a day.
  Interventions: Drug: Antroquinonol

INTERVENTIONS:
Drug: Antroquinonol — Antroquinonol will be provided as capsules of 50 mg
  Other Names: Hocena 50mg
  Arms: Antroquinonol 100 mg PO; Antroquinonol 150 mg PO; Antroquinonol 50 mg PO
Drug: placebo — The matching placebo will be packaged as Antroquinonol with appearance identical in all aspects, however, don't have the active compound(antroquinonol)
  Arms: Antroquinonol 100 mg PO; Antroquinonol 50 mg PO; Placebo

SUMMARY:
Identified the efficacy of Antroquinonol (Hocena 50mg) in triglyceride, lipid-lowering and fatty liver.

DETAILED DESCRIPTION:
The primary efficacy objective is to demonstrate the reduction of triglyceride (TG) by Antroquinonol, in comparison with placebo, after 12 weeks of treatment in patients with hypercholesterolemia and hyperlipidemia. Secondary objectives include the evaluation of the effects of Antroquinonol in comparison with placebo on other lipid parameters after 12 weeks of treatment and the effects of Antroquinonol on left ventricular diastolic function, arterial stiffness and fatty liver. The safety and tolerability of Antroquinonol will be monitored as well.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of either sex 30 to 75 years of age, inclusive, with a diagnosis of nonfamilial hypercholesterolemia or mixed hyperlipidemia as one of the following:

   * TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL
   * TG between 150 mg/dL and 500 mg/dL and LDL-C > 130 mg/dL);
2. Subject must be free of any clinically significant disease, other than nonfamilial hypercholesterolemia or mixed hyperlipidemia that would knowingly interfere with study evaluations;
3. A wash-out period of 2 weeks will be applied to patients prior treated with lipid-lowering medication;
4. Subject must be willing to adhere to protocol requirements, and provide written informed consent;
5. Female of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation.

Exclusion Criteria:

1. Patients with secondary dyslipidemia caused by diabetes mellitus, hypothyroidism, obstructive liver disease, chronic renal failure or drugs which can increase LDL-C level (e.g. retinoids, cyclosporine A and phenothiazines) or decrease HDL-C level (e.g. progestins, androgens, β-blockers, probucol and anabolic steroid)
2. Patients with lifestyle that may interfere treatment efficacy, such as alcoholism or drinking habits more than 3 times per week, late dinner, late night supper, frequent oversea business traveler, frequent social gathering, and patients who cannot anticipate a diet control and lifestyle changes;
3. Patients with diabetes or history of coronary artery disease (has had myocardial infarction, cardiac intervention, cerebrovascular accident/stroke or transient ischemic attack less than 6 months prior to Visit 1);
4. Patients with hypertension that is uncontrolled defined as 2 consecutive measurements of sitting blood pressure of systolic >140 mmHg or diastolic > 90 mmHg at Visit 1;
5. Patient has a known hypersensitivity to Antroquinonol or related compounds;
6. Patient with uncontrolled intercurrent illness including, but not limited to, acute decompensated HF (exacerbation of chronic HF manifested by signs and symptoms that may require IV therapy), right heart failure due to severe pulmonary disease, diagnosed peripartum or chemotherapy induced cardiomyopathy within the 12 months prior to visit 1, or psychiatric illness/social situations that would limit compliance with study requirements;
7. Patients with a history of heart transplant or who are on a transplant list or with left ventricular assistance device (LVAD device);
8. Patients with documented ventricular arrhythmia with syncopal episodes within the past 3 months prior to visit 1 that remained untreated;
9. Patients with confirmed severe primary pulmonary, renal (eGFR<30 ml/min/1.73 m2) or hepatic (Child-Pugh B/C classification) disease;
10. Patients who can't stop current lipid lowering drug treatments based on investigator's judgement;
11. Patients with any malignancy, treated or untreated, within the past 5 years of Visit 1 whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin or carcinoma in situ of the cervix;
12. Female patient during pregnancy, lactation or breastfeeding;
13. Patient has any other life-threatening complications;
14. Patient who is considered unreliable as to medication compliance or adherence to scheduled appointments, or inappropriate for inclusion determined by the investigators;
15. Any other reasons addressed by the investigators.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-05; Primary Completion 2018-09-27 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Tien Chiang, M.D., Principal Investigator — National Taiwan University Hopspital
Locations (6):
- Taiwan (6):
  - Chang Gung Memorial Hospital, Linkou branch, New Taipei City
  - Far Eastern Memorial Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-center, phase II, prospective, double blind, randomized, placebo-controlled trial, recruiting from 23-Jun-2016 to 30-Aug-2018 6 sites are NTUniversity Hospital; CMU Hospital; NCKU Hospital; Taipei VG Hospital; FEM Hospital; CGM Hospital, Linkou branch;
Pre-assignment Details: total treatment period: 16 weeks including a 2-week screening visit, a 12-week study treatment, and a 2-week follow-up
Groups:
- Placebo: Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (Placebo) 3 capsules once a day.
  placebo: The matching placebo will be packaged as Antroquinonol with appearance identical in all aspects, however, don't have the active compound(antroquinonol)
- Antroquinonol 50 mg PO: Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (1 capsule of antroquinnonol 50mg and 2 capsules of Placebo) 3 capsules once a day.
  Antroquinonol: Antroquinonol will be provided as capsules of 50 mg
- Antroquinonol 100 mg PO: Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (2 capsules of antroquinnonol 50mg and 1 capsule of Placebo) 3 capsules once a day.
  Antroquinonol: Antroquinonol will be provided as capsules of 50 mg
- Antroquinonol 150 mg PO: Subjects with screening central laboratory with a diagnosis of primary hypercholesterolemia (nonfamilial) or mixed hyperlipidemia (TG between 150 mg/dL and 500 mg/dL, and cholesterol between 160 mg/dL and 250 mg/dL or LDL-C > 130 mg/dL ) who meet inclusion/exclusion criteria will be randomized to 4 groups patient will take (antroquinnonol 50mg ) 3 capsules once a day.
  Antroquinonol: Antroquinonol will be provided as capsules of 50 mg
Period: Overall Study
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO
Started | 30 | 30 | 30 | 30
Completed | 28 | 28 | 24 | 20
Not Completed | 2 | 2 | 6 | 10
Not completed — Adverse Event | 2 | 1 | 4 | 8
Not completed — Physician Decision | 0 | 1 | 1 | 1
Not completed — Use of prohibited medication | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO | Total
Number analyzed (Participants) | 30 | 30 | 30 | 30 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.2 (15.12) | 53.3 (13.18) | 48.9 (10.32) | 52.5 (9.98) | 50.70 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 5 | 8 | 35
  Male | 18 | 20 | 25 | 22 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 30 | 30 | 30 | 30 | 120
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 30 | 30 | 30 | 30 | 120
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.71) | 27.2 (3.80) | 28.4 (5.41) | 26.8 (3.72) | 27.68 (4.36)

OUTCOME MEASURES:

1. Primary Outcome: TG Change (mg/dL )
Description: value at 12 weeks minus value at baseline
Time Frame: 12 weeks
Population: Per-protocol population
Measure: Median (95% Confidence Interval); unit: percentage of change
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO
Number analyzed (Participants) | 28 | 28 | 22 | 20
percentage of change | -9.2 [-17.97 to 12.20] | 14.6 [3.48 to 40.8] | -4.2 [-15.68 to 15.80] | -1.3 [-13.01 to 15.17]

2. Secondary Outcome: LDL& HDL (mg/dL)
Description: value at 12 weeks minus value at baseline of PP pupulation in HDL/LDL ratio.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO
Number analyzed (Participants) | 28 | 28 | 22 | 20
percentage of change | 2.4 (21.73) | 5.1 (23.02) | -1.1 (15.51) | 0.3 (13.98)

3. Secondary Outcome: Non-invasive Arterial Stiffness Measurement
Description: To evaluate the effect of Antroquinonol via a non-invasive arterial stiffness measurement.
Time Frame: 12 weeks
Population: Per-protocol population
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO
Number analyzed (Participants) | 28 | 28 | 22 | 20
percentage of change | 3.1 (9.58) | 0.0 (13.80) | -3.3 (10.38) | 2.8 (9.84)

4. Secondary Outcome: Fatty Liver
Description: To evaluate the recover fatty liver effect of Antroquinonol on patients who with fatty liver by Investigator
Time Frame: 12 weeks
Population: Only Per-protocol population subjects with abnormal liver attenuation at baseline subjected to follow-up after 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO
Number analyzed (Participants) | 15 | 13 | 12 | 11
Participants | 0 | 4 | 1 | 1

ADVERSE EVENTS:
Time Frame: 16 weeks start from Screening visit to follow up visit. The mean duration of dosing was 81.4 days in the placebo group, 81.3 days in the antroquinonol 50 mg group, 75.6 days in the antroquinonol 100 mg group, and 65.0 days in the antroquinonol 150 mg group.
Description: there are few patients had more than one AE during the study
Arm/Group | Placebo | Antroquinonol 50 mg PO | Antroquinonol 100 mg PO | Antroquinonol 150 mg PO
All-Cause Mortality (participants affected / at risk) | 8/14 | 8/13 | 12/19 | 17/18
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 1/19 | 0/18
Other Adverse Events (participants affected / at risk) | 8/14 | 8/13 | 12/19 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Antroquinonol 50 mg PO (N=13) | Antroquinonol 100 mg PO (N=19) | Antroquinonol 150 mg PO (N=18)
ureterolithiasis and urinary tract disorder (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — one patient has two SAEs: ureterolithiasis and urinary tract disorder. Both are not related to Antroquinonol
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=14) | Antroquinonol 50 mg PO (N=13) | Antroquinonol 100 mg PO (N=19) | Antroquinonol 150 mg PO (N=18)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 8 (8) | 9 (9) | 13 (13)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Additional study with larger sample size is warranted to confirm antroquinonol in treating hyperlipidemia, arterial stiffness, and fatty liver.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/28/NCT02719028/SAP_000.pdf
  • Study Protocol (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/28/NCT02719028/Prot_001.pdf